CLINICAL TRIAL: NCT06926179
Title: Safety, Efficacy, and Survival Outcomes of Neoadjuvant/Induction Immunotherapy in Surgical and Radiotherapeutic Management of Non-Small Cell Lung Cancer: A Multicenter Real-World Study
Brief Title: Safety, Efficacy, and Survival Outcomes of Neoadjuvant/Induction Immunotherapy in Surgical and Radiotherapeutic Management of Non-Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wu Nan, Professor, Peking University Cancer Hospital & Institute
Other Study IDs: 10412
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer (NSCLC); Neoadjuvant Immunotherapy; Radiotherapy; Lung Surgery
Keywords: lung cancer; neoadjuvant immunotherapy; real-world study; radiotherapy; thoracic surgery
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: neoadjuvant immunotherapy — Patients in the cohort received neoadjuvant immune checkpoint inhibitors (ICIs), including PD-1/PD-L1 inhibitors, as part of routine clinical care. The specific regimens included monotherapy or combination with chemotherapy. The agents used may include nivolumab, camrelizumab, sintilimab, atezolizumab, or others.
  This is a retrospective observational study. All interventions (neoadjuvant immunotherapy ± chemotherapy, surgery, or other treatments) were determined by treating physicians as part of standard care. The study aims to evaluate perioperative and survival outcomes across different treatment paths in real-world clinical settings.

SUMMARY:
This multicenter retrospective real-world study aims to evaluate the safety, efficacy and survival outcomes of neoadjuvant/induction immunotherapy in patients with non-small cell lung cancer (NSCLC). The study covers diverse treatment pathways, including surgery, definitive radiotherapy, and non-surgical strategies. It addresses gaps in existing trials by establishing a comprehensive cohort spanning neoadjuvant/induction therapy, perioperative management, and follow-up, providing real-world evidence to support treatment decisions in both operable and inoperable cases.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related deaths in both China and the world. In recent years, neoadjuvant immunotherapy has achieved breakthrough advancements in the treatment of non-small cell lung cancer (NSCLC). Evidence from multiple Phase III randomized controlled trials (RCTs), such as CheckMate 816, KEYNOTE-671, and AEGEAN, has demonstrated clear benefits of this therapy in improving survival. However, these studies exhibited several limitations: first, stringent selection criteria resulting in limited heterogeneity among participants challenge the generalizability of their conclusions; Second, some studies and clinical observations have preliminarily suggested that neoadjuvant immunotherapy may increase technical surgical difficulty; however, large-sample, real-world data on its perioperative safety remain limited; third, clinical practice involves numerous borderline resectable and unresectable cases, leading to highly complex treatment decisions (such as timing of surgical intervention after conversion therapy, radiotherapy strategies, etc.), with none of the existing guidelines reach clear consensus.

This study employs a multicenter real-world design, establishing a retrospective cohort covering from neoadjuvant/induction therapy period to the surveillance period. It evaluates the safety, efficacy, and survival outcomes of neoadjuvant/induction immunotherapy across diverse treatment strategies including both surgery and radiotherapy, providing real-world evidence to inform clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed non-small cell lung cancer (NSCLC), regardless of the presence of EGFR or ALK sensitive driver gene mutations;
2. Clinical staging of IA-IIIC according to the AJCC 8th Edition before neoadjuvant treatment;
3. Received at least one cycle of neoadjuvant immunotherapy (with or without chemotherapy);
4. Assessed as resectable or potentially resectable by surgical experts prior to treatment.

Exclusion Criteria:

1. Confirmed M1 disease;
2. History of previous lung malignancy or other metastatic malignant tumors;
3. Participation in other randomized controlled trials involving neoadjuvant treatment;
4. Significant missing clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include real-world patients diagnosed with stage IA-IIIC non-small cell lung cancer (NSCLC) who received at least one cycle of neoadjuvant immunotherapy (with or without chemotherapy). According to surgical evaluation, patients eligible for inclusion were assessed as either resectable or potentially resectable before treatment. Subsequent treatment following the neoadjuvant therapy may include surgical resection, radiotherapy, or non-localized therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Technical Dissection Difficulty (TDD) Rate | During the radical surgery (Day 0 of surgery)
  Defined as the intraoperative presence of fibrosis and/or tight adhesion between lymph nodes and surrounding structures around the hilar and fissure. TDD is considered present if either fibrosis or significant adhesion is noted, potentially increasing surgical complexity. Surgical difficulty is assessed based on operative reports and predefined intraoperative criteria, as documented by the operating surgeon.
Disease-Free Survival (DFS) | From the date of radical surgery to the date of disease recurrence, progression, death, or last follow-up, up to 5 years.
  Defined as the time from the date of radical surgery to the first occurrence of disease recurrence, progression, or death from any cause. Patients without an event will be censored at the date of the last follow-up. Disease status is determined through radiological, pathological, or clinical assessment as documented during follow-up.

SECONDARY OUTCOMES:
Postoperative Complications Incidence (Clavien- Dindo ≥ III) | Within 30 days after surgery
  Defined as the proportion of patients experiencing postoperative complications graded as Clavien-Dindo classification grade III or higher within 30 days after radical surgery. Complication data are collected from postoperative records, discharge summaries, and follow-up documentation.
Treatment-Related Adverse Events (TRAEs) Incidence (CTCAE Grade ≥ 3) | From the start of neoadjuvant or induction therapy to 90 days after the initiation of definitive local treatment (surgery or radiotherapy).
  The incidence of treatment-related adverse events (TRAEs) graded ≥3 according to the Common Terminology Criteria for Adverse Events (CTCAE), v5.0, occurring during the neoadjuvant/induction phase and within 90 days following the initiation of definitive local therapy (surgery or radiotherapy). TRAEs are assessed based on clinical presentation, laboratory findings, imaging results, and physician judgment, with causality reviewed by the research team.
Immune-Related Adverse Events (irAEs) Incidence | From the start of neoadjuvant or induction therapy to 90 days after the initiation of definitive local treatment (surgery or radiotherapy).
  Defined as the incidence of immune-related adverse events (irAEs) occurring from the start of neoadjuvant immunotherapy until 90 days after radical surgery or the initiation of definitive radiotherapy, whichever applies. irAEs are adverse events potentially attributable to immune checkpoint inhibitors and may involve organs such as the lung, liver, skin, or endocrine system. Events are graded according to CTCAE v5.0, and diagnosis is based on clinical presentation, laboratory/imaging findings, and expert clinical judgment.
Progression-Free Survival (PFS) | From the start of neoadjuvant immunotherapy to the date of disease progression, death, or last follow-up, up to 5 years.
  Defined as the time from the initiation of neoadjuvant immunotherapy to the first documented disease progression or death from any cause, whichever occurs first. Disease progression includes local recurrence, regional relapse, distant metastasis, or any clinically or radiologically confirmed progression. Patients without an event will be censored at the date of the last follow-up.
Overall Survival (OS) | From the date of treatment initiation to death from any cause or last follow-up, up to 5 years
  Defined as the time from the initiation of neoadjuvant therapy to death from any cause. For patients who remain alive at the end of follow-up, OS will be censored at the date of the last known contact. Survival status is confirmed through electronic medical records, follow-up visits, or telephonic interviews. OS is measured in days and analyzed using time-to-event methods.
Conversion Rate to Thoracotomy | During the radical surgery (Day 0)
  Defined as the proportion of patients initially planned for video-assisted thoracoscopic surgery (VATS) who required unplanned conversion to open thoracotomy during radical resection. Conversion events and their intraoperative causes will be extracted from operative records and confirmed by surgical documentation. The outcome reflects intraoperative difficulty and is used as a surrogate marker of surgical complexity.
Operative Time (minutes) | During the radical surgery (Day 0)
  Defined as the total operative time, measured in minutes, from the initial skin incision to the completion of skin closure during radical lung resection. Time data are extracted from intraoperative anesthesia or surgical records. Operative time is used as a continuous variable and may reflect the technical complexity of surgery.
pathologic Complete Response (pCR) Rate | At the time of postoperative pathological assessment
  Defined as the proportion of patients achieving a pathologic complete response (pCR), which is characterized by the absence of any viable tumor cells in the resected primary tumor and all sampled regional lymph nodes (ypT0N0), as confirmed by postoperative pathological examination. Pathologic assessments are conducted by experienced thoracic pathologists according to standardized criteria.
Major Pathologic Response (MPR) Rate | At the time of postoperative pathological assessment
  Defined as the proportion of patients achieving a major pathologic response (MPR), characterized by ≤10% residual viable tumor cells in the resected primary tumor specimen after neoadjuvant therapy, regardless of lymph node status. The percentage of residual tumor is assessed by experienced thoracic pathologists according to standardized pathological evaluation protocols.
Number of Dissected Lymph Nodes (N1, N2) | During radical surgery (Day 0)
  Defined as the total number of lymph nodes dissected and pathologically examined from N1 and N2 stations during radical lung cancer resection. The counts are recorded separately for N1 and N2 regions based on operative and pathological reports. This outcome reflects the extent of mediastinal and hilar lymphadenectomy and may serve as an indicator of surgical thoroughness and potential prognostic value.
Number of Dissected Lymph Node Stations (N1, N2) | During radical surgery (Day 0)
  Defined as the number of lymph node stations sampled or dissected from the N1 and N2 regions during radical lung cancer surgery. The count is recorded separately for N1 and N2 stations based on operative and pathological reports. This measure reflects the anatomical extent of lymphadenectomy and is used to evaluate surgical thoroughness and adherence to oncologic guidelines.
Reduction Rate of Surgical Resection Extent | During the radical surgery (Day 0 of surgery)
  Among patients whose anticipated surgical resection before neoadjuvant immunotherapy involved more than one pulmonary lobe, this outcome measures the proportion whose actual surgical resection was less extensive than originally planned. The anticipated extent is based on pre-treatment multidisciplinary evaluations, including imaging and bronchoscopy.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Inner Mongolia Hospital of Peking University Cancer Hospital, Hohhot, Inner Mongolia
  - The Third Affliated Hospital of Kunming Medical University, Kunming, Yunnan